CLINICAL TRIAL: NCT05667376
Title: Efficacy of Curcumin Gel as an Adjunct to Scaling and Root Planing on Salivary Procalcitonin Level in the Treatment of Periodontitis Patients: Randomized Controlled Clinical Trial
Brief Title: Efficacy of Curcumin Gel Combined With Non-surgical Periodontal Therapy on Salivary Procalcitonin Level in the Treatment of Periodontitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reham abdelfatah (Other)
Responsible Party: Sponsor-Investigator, Reham abdelfatah, BDS, Clinical demonstrator, Oral Medicine, Periodontology, Diagnosis, and Oral Radiology Department,, Mansoura University
Organization: Mansoura University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A01031120
Record Dates: First submitted 2022-10-03; First posted 2022-12-28 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: patients (n=70) were selected from the Department of Oral Medicine and Periodontology, Faculty of Dentistry, Mansoura University, sixteen patients (n=16) were excluded as eight patients (n=6) weren't met the inclusion criteria and the other eight patients (n= 6) declined to participate with (n=4) were excluded due to pregnancy and lactation. The participants fifty -four patients were classified into three groups: group I (healthy individuals), group II (SRP group), and group III (curcumin gel group). Patients in group II and group III included patients with stage II grade A periodontitis. Patients in group II were treated with SRP only while in group III curcumin gel was applied weekly for four weeks after SRP had been completed.
Masking Description: The patients with periodontitis groups were randomly selected into either group II or III using the coin toss method. Hence the study groups were classified into three groups as follows, group I (negative control group): eighteen subjects with clinically healthy gingiva were selected to participate in the study as a reference group, and group II (positive control group): eighteen patients with periodontitis (stage II grade A) were selected and treated with non-surgical periodontal therapy (SRP) only, and group III (study group): eighteen patients with periodontitis (stage II grade A) were selected and treated with SRP followed by curcumin gel application
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Other): Study group treated with curcumin gel
  Interventions: Other: Local drug delivery; Drug: curcumin gel

INTERVENTIONS:
Other: Local drug delivery — Local application of curcumin gel into the periodontal pocket
Drug: curcumin gel — curcumin gel

SUMMARY:
Objectives: To evaluate the efficacy of curcumin gel as an adjunct to scaling and root planing (SRP) on the salivary procalcitonin level in the treatment of periodontitis.

Materials and methods: seventy patients (n=70) were selected from the Department of Oral Medicine and Periodontology, Faculty of Dentistry, Mansoura University, sixteen patients (n=16) were excluded as eight patients (n=8) weren't met the inclusion criteria, and other eight patients were divided into (n= 4) declined to participate with (n=4) were excluded due to pregnancy and lactation. The participants fifty -four patients were classified into three groups: group I (healthy individuals), group II (SRP group), and group III (curcumin gel group). Patients in groups II and III included stage II grade A periodontitis. Patients in group II were treated with SRP only while in group III curcumin gel was applied weekly for four weeks after SRP had been completed. Clinical indices (plaque index (PI), gingival index (GI), clinical attachment level (CAL), and probing depth (PD)) and saliva samples for procalcitonin (PCT) assessment using an enzyme-linked immunosorbent assay (ELISA) test were collected and measured at baseline and again after six weeks.

DETAILED DESCRIPTION:
Study population The randomized controlled clinical trial included fifty-four participants selected from the Department of Oral Medicine and Periodontology Outpatient Clinic, Faculty of Dentistry, Mansoura University from January 2021 to May 2021. Thirty-six patients with periodontitis (stage II grade A) and eighteen healthy volunteers (negative control group) participated in the study.

A. Inclusion criteria for patient selection: The selected patients included:

1. Participants of both sexes between the ages of thirty to fifty -five years old
2. Participants with periodontitis (stage II grade A with PD of 3-5 mm and CAL of 3-4mm).

B. Exclusion criteria included:

1. Participants with known systemic diseases
2. Pregnant and lactating participants.
3. Tobacco (smoking/chewing).
4. History of antibiotic and periodontal therapy in the last 3 months.
5. Participants who weren't compliant with oral hygiene procedures.

Study Design: The selected patients will be divided into 3 groups:

Group 1 (study group): patients are to be treated with turmeric gel as an adjunct to Scaling and root planing.

Group 2 (positive control group): patients are to be treated with only Scaling and root planing.

Group 3 (negative control group): patients with clinically healthy gingiva.

3) Periodontal Assessment:

All these measurements will be assessed :

1. Plaque Index according to Silness P. Loe H 1964.
2. Gingival Bleeding Index according to Ainamo & Bay 1975.
3. Probing pocket depth (PPD) is measured from the free gingival margin to the base of the pocket.
4. Clinical attachment level (CAL) is measured from the cement enamel junction to the base of the pocket.

For all periodontitis patients, the Clinical assessment will be performed at baseline and 45 days after periodontal treatment ( either Scaling, root planning, and injection of gel or Scaling and root planning alone ).

This study was conducted following guidelines regulating research work on human subjects of the Faculty of Dentistry, Mansoura University, and the study protocol was reviewed and approved by the Research Ethics Committee of the Faculty of Dentistry, Mansoura University, Egypt. (Number: A01031120).

Sample size calculation Sample size calculation was based on mean superoxide dismutase (SOD) after treatment between the study and control group retrieved from a previous study (Elavarasu et al., 2016). Using G*power version 3.0.10 to calculate sample size based on the effect size of 0.828, 2-tailed test, α error =0.05, d power = 90.0% the total calculated sample size was 18 in each group at least.

Pretreatment period Participants were informed about the purpose of the study and screened for eligibility. They also were informed about the treatment received and the steps done, including non-surgical treatment and gel application with the associated risks, possible effects, and other treatment options available. The participants understood this explanation in broad terms according to the rules of the ethical committee of the Faculty of Dentistry, Mansoura University. Additionally, they acknowledged that they would be required to attend the periodic recall visits and that they are legally competent to give written informed consent before performing any required steps.

Randomization and study groups The patients with periodontitis groups were randomly selected into either group II or III using the coin toss method. Hence the study groups were classified into three groups as follows, group I (negative control group): eighteen subjects with clinically healthy gingiva were selected to participate in the study as a reference group, and group II (positive control group): eighteen patients with periodontitis (stage II grade A) were selected and treated with non-surgical periodontal therapy (SRP) only, and group III (study group): eighteen patients with periodontitis (stage II grade A) were selected and treated with SRP followed by curcumin gel application.

Saliva sample collection:

Saliva sample collection was accomplished using the swabbing method. It was performed by introducing a cotton pad into the mouth at the orifices of major salivary glands. The subjects were asked to chew the cotton pad to get soaked in the saliva. The saliva-soaked pad was removed and placed in a sterile test tube (sterile Eppendorf tube) and centrifuged at 3000 rounds per minute (RPM) for approximately 10 minutes and then kept frozen at -20°c till the time of analysis.

Procedures for curcumin gel preparation:

Curcumin Gel Preparation: The gel will be prepared in the Department of Pharmacology, Faculty of Pharmacy, Mansoura University. Preparation of 2% curcumin gel by simple dispersion method as shown: Formula to prepare 2%curcumin gel Ingredients Quantity Carpacol 2 gm Polymer (HPMC) 2 gm Curcumin 5 ml Propylene glycol 0.2 ml Sodium benzoate q.s Triethanolamine q.s. to make 100 ml Distilled water 2g

(HPMC =hydroxy propyl methyl cellulose ; q.s.=quantity sufficient) Carbopol 940 will be soaked in purified water containing 0.2% w/v sodium benzoate overnight. Using tissue homogenizer hydroxypropyl methylcellulose (HPMC) solution will be mixed in propylene glycol. 0. 2 mg of curcumin (Sigma, St. Lo, USA) will be transferred into HPMC solution and homogenized. This drug solution will be transferred to a carbopol solution and homogenized. Triethanolamine will be added in a quantity sufficient (q.s.) to neutralize the pH. Then, distilled water will be added to make q.s. to 100 ml. The gel will be stored at ambient temperature. The prepared gel will be tested for microbial growth by incubation for 24 hours. If no microbial growth will be observed, the final preparation will then be transferred into glass containers and will be stored in the refrigerator (temperature ranging from 2-10°C and 80-85% humidity)

SRP procedures:

At the beginning of treatment, the periodontitis patients were treated with SRP using both special tipped ultrasonic scalers and manual Gracey curettes until a smooth tooth/root surface was achieved. The SRP procedure was repeated once again (if necessary) and instructions were given to the patients to maintain good oral hygiene measures during the treatment period. Brushing and flossing techniques were taught to all participants using patient education videos and demonstrated on study models. No antibiotics or mouthwashes were prescribed during treatment. All patients were recalled weekly during the study period (which was carried out for six weeks) for reinforcement of oral hygiene measures and curcumin gel application inside the only selected periodontal pockets of group III as it was applied weekly for four weeks after completing SRP.

Curcumin Gel Application:

Following SRP procedures, only selected periodontal pockets (pockets diagnosed with stage II grade A, PD of 3-5 mm, and CAL of 3-4mm) within group III were delivered with 2% curcumin gel sub-gingivally using a disposable 2 ml syringe with a blunt needle (bent 130° at the shank). The application of gel was initiated from the base of the pocket to ensure the gel reached the whole pocket depth. This was accomplished by a plastic syringe with a flexible metal needle with a large gauge (similar to those used for acid etchant application).

This procedure continued until the pocket was filled. Care was taken to apply the gel without traumatizing or damaging the periodontal tissues. After insertion of the curcumin gel, the region was secured with a cotton pack, and the patients were advised not to eat or drink for at least two hours following gel administration. They were also advised not to brush the treated areas or floss /use interproximal cleaning devices for at least twelve hours postoperatively and to avoid eating hard and abrasive foods that could traumatize the gingiva. The treatment was followed-up by weekly recalls after gel application for reinforcement of oral hygiene measurements and subsequent gel reapplication. The curcumin gel was applied weekly for four weeks after completing SRP.

Periodontal measurements ( plaque Index (PI ), gingival index (GI), probing depth (PD), and clinical attachment level (CAL) were recorded at baseline for all groups and again six weeks after periodontal treatment for both group II and group III using a periodontal probe as most studies outcomes were assessed based on either short-term effects (studies with a 2-weeks follow-up, acceptability range ±3 days) or long-term effects (studies with a 4-weeks follow-up, acceptability range ±3 days). Measurements were done by a blinded single examiner (SE) who did not know the identity of the groups in which patients were included.

Intra-examiner reliability To achieve intra- examiner calibration, periodontal measurements of 10 patients were performed twice within 2 days before randomized clinical trial (RCT) conduction. Calibration was approved when measurements of PD and CAL in the two instances were within a 1 mm variance in more than 90% of all measurements.

Laboratory assessment of PCT level The salivary samples were collected from all participants at baseline and once more from both group II and group III after six weeks. The samples were kept in sterile Eppendorf tubes, centrifuged at 3000 RPM for approximately 10 minutes, and frozen at -20°c until the time of analysis by ELISA test to assess salivary PCT (according to manufacturer instructions).

Statistical Assessment:

Data will be analyzed using SPSS (statistical package for social sciences) version 22. Qualitative data will be presented as numbers and percentages, Quantitative data will be tested for normality by the Shapiro-Wilk test and then described as mean and standard deviation for normally distributed data and median and range for non-normally distributed. The appropriate statistical test will be applied according to the data type with the following suggested tests: Chi-Square for categorical variable. One Way ANOVA and Kruskal-Wallis tests U test for continuous variables. Repeated Measures ANOVA and Freidman tests for comparing pre, post, and follow-up readings. Pearson and spearman correlation will be used to correlate between continuous variables

ELIGIBILITY:
Inclusion Criteria:

* inclusion criteria were participants of both sexes, between the ages of thirty and fifty -five years old with periodontitis (stage II grade A).

Exclusion Criteria:

* exclusion criteria involved participants with known systemic diseases, pregnant and lactating patients, tobacco users (smoking /chewing), history of antibiotic and periodontal therapy in the last three months, and participants who weren't compliant with oral hygiene procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth reduction | Six weeks
  Clinical attachment level gain

CONTACTS AND LOCATIONS:
Overall Officials: Reham A Abdel-Fatah, Principal Investigator — Mansoura university Faculty of dentistry
Locations (1):
- Reham Ahmed Abdel-Fatah, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abdel-Fatah R, Mowafey B, Baiomy A, Elmeadawy S. Efficacy of curcumin gel as an adjunct to scaling and root planing on salivary procalcitonin level in the treatment of patients with chronic periodontitis: a randomized controlled clinical trial. BMC Oral Health. 2023 Nov 19;23(1):883. doi: 10.1186/s12903-023-03512-y. PMID 37981665